CLINICAL TRIAL: NCT04011085
Title: Tw HER2 Positive Breast Cancer Productivity & Utility Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taiwan Epidemiology Association (Other)
Responsible Party: Sponsor
Other Study IDs: ML40952
Record Dates: First submitted 2019-04-10; First posted 2019-07-08 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: HER2-positive Breast Cancer
Keywords: HER2-positive Breast Cancer; work productivity; health-related quality of life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group1: Patients currently undergoing treatment for early breast cancer (either targeted HER2 therapy and chemotherapy OR targeted HER therapy alone)
- Group2: Patients with early breast cancer who have completed treatment and are in disease-free survival (i.e. no longer receiving locoregional treatment, chemotherapy or targeted HER2 therapy; patients may still be receiving hormone therapy)
- Group3: Patients receiving treatment for metastatic breast cancer

SUMMARY:
Breast cancer ranks top 4 Taiwan mortality cause in 2016 and the incidence rate has been increasing. Since advances in screening and treatment over last decades, disease-free survival in HER2 positive breast cancer improved and relapse rates decrease as well. While health-related quality of life (HRQoL) and productivity benefit is not currently formally assessed by Taiwan Health Technology Agency (HTA) in Taiwan, the value of therapy in terms of a wider societal benefit is a critical factor which is increasingly being considered as part of the overall assessment of the value of a new medicine.

Sort of productivity study in cancer is lack of in Taiwan. Referenced Roche UK team published comprehensive productivity studies1 Taiwan Epidemiology Association wants to initiate study to understand holistic value in each stage of breast cancer and quantify the value of new drug to support HTA assessment.

The data will be collected through study, and adapt to cost-effectiveness model for future reimbursement submission.

DETAILED DESCRIPTION:
Breast cancer ranks top 4 Taiwan mortality cause in 2016 and the incidence rate has been increasing. Since advances in screening and treatment over last decades, disease-free survival in HER2 positive breast cancer improved and relapse rates decrease as well. While health-related quality of life (HRQoL) and productivity benefit is not currently formally assessed by Taiwan Health Technology Agency (HTA) in Taiwan, the value of therapy in terms of a wider societal benefit is a critical factor which is increasingly being considered as part of the overall assessment of the value of a new medicine.

Sort of productivity study in cancer is lack of in Taiwan. Referenced Roche UK team published comprehensive productivity studies1 Taiwan Epidemiology Association wants to initiate study to understand holistic value in each stage of breast cancer and quantify the value of new drug to support HTA assessment.

The data will be collected through study, and adapt to cost-effectiveness model for future reimbursement submission.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or over;
* Diagnosed with early stage or metastatic (Stage IV) HER2-positive breast cancer (confirmed by the study site physician). [HER2-positive is defined as IHC3+ and/or ISH≥2.0]
* eBC patients should have received at least 2 cycles of adjuvant anti-cancer therapy following surgery at time of interview; metastasis breast cancer (mBC) patients should have received at least 1 cycle of treatment for their metastatic disease at time of interview.
* Able to provide written, informed consent.

Exclusion Criteria:

* Patients with ECOG performance status (PS) ≥3
* Unwilling or unable to provide written, informed consent
* Unable to complete written quality of life questionnaires

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HER2 POSITIVE BREAST CANCER
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-12-24 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Work Productivity and Activity Impairment | 1 year
  • Percent work time missed due to health: Hours missed due to health problems/(Hours missed due to health problems+ Hours actually worked)
  • Percent impairment while working due to health: Degree health affected productivity while working/10
  • Percent overall work impairment due to health: Hours missed due to health problems/(Hours missed due to health problems+ Hours actually worked)+[(1-( hours missed due to health problems/( hours missed due to health problems+ hours actually worked)))x(degree health affected productivity while working/10)]
  • Percent activity impairment due to health: Degree health affected regular activities/10

SECONDARY OUTCOMES:
EQ-5D-5L | 1 year
  The descriptive system of EQ-5D-5L comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), and each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems.
EQ Visual Analogue scale (EQ VAS) | 1 year
  The EQ VAS records the respondent's self-rated health on a visual analogue scale.
Functional Assessment of Cancer Therapy-Breast Cancer (FACT-B) | 1 year
  the FACT-B consists of the following subscales: physical well-being (PWB), functional well-being (FWB), emotional well-being (EWB), social/family well-being (SWB), and breast cancer-specific concerns (BCS). A total FACT-B score is calculated by summing the subscales. The instrument has a total of 41 items asking respondents to rate how true each statement is for the last 7 days. Response scales range from 0 (not at all) to 4 (very much).
Demographics | 1 year
  age, gender, height, weight, marital status, education level, employment status, monthly household income, and family history of breast cancer
Site of survey administration | 1 year
  north, central and south

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Hung Lin, Ph.D, Study Chair — National Taiwan University Hospital; Liang-Chih Liu, Ph.D, Study Chair — China Medical University Hospital; Ming-Feng Hou, M.D., Study Chair — Kaohsiung Medical University
Locations (1):
- National Taiwan University hospital, Taipei, Taiwan